CLINICAL TRIAL: NCT07325760
Title: 1. Translating MY-MINDD Into Practice: Retort Meal Interventions to Improve Muscle Health, Nutritional Status, and Food Security Among Malaysian Older Adults 2. Effectiveness of ReMIND Diet- Based Retort Meal Intervention on Cognitive Frailty in Low-Income Malaysian Older Adults: A Cluster Randomised Controlled Trial
Brief Title: Effectiveness of a ReMIND Diet Intervention on Sarcopenia, Cognitive Frailty and Nutritional Status in Older Adults
Acronym: ReMIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: United Nations (Other)
Responsible Party: Principal Investigator, Chan Yoke Mun, Prof. Dr. Chan Yoke Mun, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JKEUPM-2025-383
Record Dates: First submitted 2025-11-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Cognitive Frailty; Nutritional Interventions
Keywords: older adults; sarcopenia; cognitive; cognitive frailty; malnutrition; mind diet; my-mindd; nutrition intervention
MeSH Terms: conditions — Sarcopenia; Malnutrition

STUDY DESIGN:
Intervention Model Description: A 12-week, two-arm, cluster randomized controlled trial, quantitative study.
  This study adopts an experimental design, specifically a 12-week, two-arm, cluster randomized controlled trial (RCT). Cluster allocation will be determined by simple randomization. Between the two comparable housing clusters, PPR Seri Alam Fasa 2 and PA Loke Yew, the intervention and control groups will be assigned by drawing lots. PPR Seri Alam Fasa 2 was randomly designated as the intervention cluster, while PPA Loke Yew served as the control cluster. Under this randomization process, eligible participants from PPR Seri Alam Fasa 2 will receive the retort meals through the MoW program for 12 weeks, while participants from PPA Loke Yew will form the control group and will only receive the retort meals after the completion of the study.
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the nutrition intervention, participants cannot be blinded to group assignment. To reduce bias, however, the researchers responsible for data entry and analysis will be blinded. Group assignments will be coded as "Group A" and "Group B" by the supervisor, and researchers will enter and analyze data without knowledge of which cluster corresponds to the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPA Loke Yew (Control Group) (No Intervention): Participants in the control group will continue with their usual daily dietary intake and routine living activities without receiving any intervention throughout the 3-month study period. However, they will be assured that they will receive the reMIND meals upon study completion, both for ethical reasons and as an appreciation for their participation and cooperation, known as wait-list control design. This post-study provision also aims to help alleviate food insecurity among participants.
  This arrangement ensures ethical equity between groups while maintaining the validity of the control condition. It may also help enhance participants' dietary awareness and motivation toward healthier eating habits in the future. Data collection for this group will occur three times, at baseline (week 1), mid-intervention (week 6), and post-intervention (week 12), mirroring the schedule of the intervention group to maintain consistency. To minimise bias, basic nutrition education will be provided.
- PPA Seri Alam Fasa 2 (Intervention Group) (Experimental): Participants in the intervention group will receive home-delivered reMIND meals for a duration of 3 months, in addition to their usual dietary intake and daily activities. The retort meals will be nutritionally balanced and portion-controlled, designed in accordance with the Recommended Nutrient Intakes (RNI) Malaysia for older adults and the MY-MINDD dietary concept. These meals are formulated to meet the nutritional requirements outlined by the MY-MINDD framework, emphasising nutrient density and cognitive health support.
  Each participant will receive two meals per day, delivered once weekly, and will be encouraged to consume the meals as part of their regular diet. All meal plans will be developed by qualified dietitians and nutritionists to ensure appropriate macronutrient and micronutrient composition, food safety, and palatability.
  At the baseline visit, participants will receive brief dietary guidance and educational materials.
  Interventions: Other: PPR Seri Alam Fasa 2 (Intervention Group)

INTERVENTIONS:
Other: PPR Seri Alam Fasa 2 (Intervention Group) — Participants in the intervention group will receive home-delivered reMIND meals for a duration of 3 months, in addition to their usual dietary intake and daily activities. The retort meals will be nutritionally balanced and portion-controlled, designed in accordance with the RNI 2017 Malaysia for older adults and the MY-MINDD dietary concept. These meals are formulated to meet the nutritional requirements outlined by the MY-MINDD framework, emphasising nutrient density and cognitive health support.
  Each participant will receive two meals per day, delivered once weekly, and will be encouraged to consume the meals as part of their regular diet. All meal plans will be developed by qualified dietitians and nutritionists to ensure appropriate macronutrient and micronutrient composition, food safety, and palatability.
  At the baseline visit, participants will receive brief dietary guidance and educational materials.
  Other Names: reMIND
  Arms: PPA Seri Alam Fasa 2 (Intervention Group)

SUMMARY:
This research is a single-blinded, 12-week, two-arm cluster randomized controlled trial to evaluate the effectiveness of a Malaysian-adapted MIND (Mediterranean-DASH Intervention for Neurodegenerative Delay) diet retort meal intervention on sarcopenia risk, cognitive frailty status, nutritional status, depression, functional ability, and food security among older adults in Malaysia. With Malaysia projected to become an aged society by 2030, addressing age-related health challenges, including cognitive frailty and sarcopenia, is a national priority. Current evidence indicates that poor diet quality and food insecurity among older adults, especially those in low-income urban communities, exacerbate these conditions. The study is grounded on the Meals on Wheels (MoW) program, which has been effective in reducing malnutrition among older populations globally but is limited in scalability due to high delivery costs. Retort meals which are shelf-stable and nutritionally balanced offer a feasible alternative for meal provision in poor urban settings. The MIND diet, originally designed to support brain health, also demonstrates benefits for muscle health and overall physical function. However, its adaptation to the Malaysian context is crucial due to cultural dietary preferences and cost barriers to certain ingredients. The intervention will recruit 70 older adults (aged 60-84 years) from Program Perumahan Rakyat (PPR) Seri Alam Fasa 2 and Perumahan Awam (PA) Loke Yew in Kuala Lumpur, classified under the B40 income group and at risk of food insecurity. The intervention group will receive retort meals designed according to the adapted MIND diet principles, while the control group will not receive intervention. Data will be collected at baseline, 6 weeks, and 12 weeks to assess outcomes in muscle health, cognitive frailty, nutritional status, depression, functional ability, food security, and cost-effectiveness. Overall, the conceptual framework provides a structured approach to understanding how the intervention contributes to improved nutritional well-being and supports the economic viability of the Meals on Wheels program. Potential confounding variables, including socioeconomic status, baseline health conditions, social support, and lifestyle factors, may also influence the outcomes. Participants will fill up a questionnaire regarding their sociodemographic characteristics, medical factors, psychological factors, lifestyle factors, food security status, functional ability, and depression status. Besides, the researcher will conduct face-to-face interviews to collect data regarding anthropometric measurements, handgrip strength, medical costs, and diet history. Statistical analyses will employ mixed-effects models to evaluate both continuous and categorical outcomes over time. The findings will generate crucial evidence on the feasibility, effectiveness, and cost-efficiency of using retort meals within MoW programs in Malaysia. Furthermore, it will inform national strategies to address food insecurity, promote healthy ageing, and reduce the burden of age-related health conditions. With Malaysia's rapidly ageing population and increasing prevalence of sarcopenia and cognitive frailty, this study has the potential to shape policy and practice by offering a sustainable, culturally tailored nutrition intervention. The evidence derived will support the scaling up of MoW programs using retort meals and contribute to long-term solutions for improving the quality of life and independence of older adults in Malaysia.

DETAILED DESCRIPTION:
Background:

Global population ageing is accelerating, with adults aged ≥60 years expected to reach 2.1 billion by 2050. Malaysia is projected to become an aged nation by 2030, when more than 15% of the population will be older adults. Ageing is associated with increased risks of chronic diseases, frailty, sarcopenia, and cognitive decline, contributing to reduced independence and quality of life. Nutrition plays a key protective role in mitigating these risks.

The MIND diet integrates principles from the Mediterranean and DASH dietary patterns and emphasizes leafy green vegetables, whole grains, legumes, nuts, fish, and limited intake of saturated fats and refined foods. Its Malaysian adaptation, MY-MINDD, incorporates culturally relevant foods, locally available fruits, soy-based products, and regionally preferred fish while excluding alcohol-based components. Previous local findings indicate that adherence to MY-MINDD is associated with improved cognitive outcomes in older adults.

Despite these benefits, poor diet quality, high reliance on eating-out patterns, and food insecurity remain prevalent among Malaysian older adults, especially among low-income urban communities. Approximately one-third of older adults in Malaysia are malnourished, and rising living costs further restrict access to nutritious foods. MoW programs offer support to food-insecure older adults but often face logistical, financial, and sustainability challenges. Integrating MY-MINDD principles into MoW through shelf-stable retort meals may enhance dietary access, improve nutritional status, and reduce risks of sarcopenia and cognitive frailty among vulnerable older adults.

Problem Statement and Rationale:

Evidence evaluating MoW programs in Malaysia remains limited, and no studies have assessed the feasibility, cost-effectiveness, or health impact of providing MIND-based retort meals within MoW delivery systems. The MIND diet has shown potential for improving diet quality, elevating neuroprotective biomarkers, and reducing risks of sarcopenia and cognitive decline; however, local implementation and evaluation remain scarce. Cultural adaptations are essential to ensure relevance in the Malaysian context.

This study addresses these evidence gaps by examining the effectiveness and cost-efficiency of integrating MY-MINDD-based retort meals into MoW programs. The investigation focuses on sarcopenia, cognitive frailty, nutritional status, depression, functional ability, and food security among economically deprived older adults.

Significance of the Study:

The intervention aligns with national guidelines emphasizing the provision of safe, nutritionally balanced, and culturally appropriate meals for vulnerable populations. The use of retort meals supports food safety, reduces logistical burdens, and enhances accessibility for older adults living in urban low-income environments. By targeting the unique challenges faced by the urban poor, such as higher food prices and limited mobility, the study contributes to national efforts to reduce food insecurity and promote healthy ageing.

Conceptual Overview:

The conceptual framework proposes that the MY-MINDD retort meal intervention will improve muscle health, cognitive frailty, nutritional status, depression, and food security. Process measures include meal satisfaction, adherence, and cost-effectiveness to assess acceptability and sustainability. Potential confounding factors include socioeconomic characteristics, baseline medical conditions, psychosocial support, and lifestyle behaviors.

Study Design:

The study utilizes a 12-week, two-arm, single-blinded, cluster randomized controlled trial. Two comparable low-income housing clusters in Kuala Lumpur (PPR Seri Alam Fasa 2 and PPA Loke Yew) serve as the randomization units. Cluster assignment is determined through simple random allocation. The intervention cluster receives MY-MINDD-based retort meals through the MoW program for 12 weeks, while the control cluster undergoes the same assessment schedule and receives the meals after study completion, known as the wait-list control. Cluster randomization is used to reduce contamination and reflect real-world MoW implementation.

Study Location:

The study is conducted in PPR Seri Alam Fasa 2 and PA Loke Yew, Kuala Lumpur. These sites have substantial populations of older adults in the B40 socioeconomic group, established community networks, and feasible distribution channels for MoW services.

Study Population and Sampling:

The target population includes Malaysian older adults aged 60-84 years residing in selected clusters and classified under the B40 income category. These individuals face higher risks of food insecurity and malnutrition. Recruitment is conducted through purposive selection of clusters and snowball sampling within each cluster. The total sample comprises 70 participants (35 per cluster).

Sample Size Justification:

A total of 70 participants is considered sufficient based on comparability with previous randomized nutrition intervention trials with similar sample sizes and measurable outcomes. The 12-week intervention is expected to produce detectable changes in nutritional and functional outcomes relevant to older adults.

Intervention Description:

The MY-MINDD diet incorporates Malaysian food culture and locally available nutrient-dense ingredients. Menu development is conducted by qualified dietitians and nutritionists to ensure compliance with dietary principles and nutrient adequacy for older adults.

Participants in the intervention group receive:

Two MY-MINDD-based retort main meals per day, five days per week (10 meals weekly) Legume-based snacks (two to three times weekly) Weekly distributions of vacuum-packed vegetables, fresh fruits, and soy milk Retort meals are produced using standardized high-temperature processing to ensure safety, extended shelf life, and nutritional preservation. Participants receive printed user guides and safety instructions on meal reheating, food handling, and emergency procedures. Weekly distribution sessions include brief feedback collection to monitor adherence, acceptability, and meal quality.

Participants in the control group receive no meals during the study period but follow identical assessment schedules. They receive MY-MINDD retort meals after completion of the study to ensure ethical fairness.

Research Instruments:

Validated and standardized instruments are used to collect data on:

Socioeconomic characteristics and medical history Diet quality (MY-MINDD scoring system) Food security (Household Food Security Survey Module (HFSSM) (USDA 6-Item version)) Depression (Geriatric depression scale -15 (GDS-15)) Anthropometry (body weight, height or arm span, waist circumference, calf circumference, body composition via Bioelectrical Impedance Analysis (BIA)) Sarcopenia (Asian Working Group for Sarcopenia (AWGS) 2019 criteria) Cognitive frailty (Montreal Cognitive Assessment (MoCA) and Fried Frailty Phenotype (FFP)) Blood biomarkers (Brain-Derived Neurotrophic Factor (BDNF)) Sun exposure indices (Sun Exposure and Protection Index (SEPI), Sun Exposure Index (SEI)) Cost-effectiveness measures (health-related costs and quality-of-life metrics)

Data Analysis:

Quantitative analyses include paired t-tests, ANOVA, chi-square tests, and logistic regression. Mixed-effects models will evaluate repeated measures across clusters and time points. Continuous variables will be analyzed using linear mixed-effects models, while categorical outcomes will be analyzed using generalized linear mixed models with random intercepts for cluster and participant.

Future Directions and Sustainability:

The intervention has potential for scalability in community-based nutrition programs for older adults. Long-term sustainability may be strengthened through collaboration with local councils, welfare departments, and food industry partners. Cost-effectiveness findings may inform policymaking, budgeting, and nationwide MoW implementation. Embedding the program within existing community support systems may enhance continuity and maximize public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian older adults aged 60 to 84 years.
* Classified under the B40 income group.
* Preferably living independently, without receiving daily meals from family members; cohabitation with other older adults is acceptable if meal support is not provided.
* Experiencing food insecurity as assessed by screening questionnaires.
* Able to provide informed consent.
* Participate in the study for the full duration.
* Able to stand without support.
* For older adults living with a spouse, preferably both partners must be eligible, willing to participate, and recruited for the study.

Exclusion Criteria:

* Individuals with diagnosed terminal illnesses (e.g., cancer, end-stage liver failure, end-stage lung disease, and severe form of heart diseases) and having medical conditions requiring specialized dietary restrictions (e.g., chronic/end-stage renal disease, severe dysphagia).
* Those with cognitive impairments or disabilities that prevent them from understanding the study procedures or providing consent.
* Participants or their spouse enrolled in other nutrition-related intervention programs during the study period.
* Those unwilling or unable to adhere to the intervention protocol.
* Bedridden
* Handicapped or amputated
* Wearing pacemaker
* Vegetarian, food allergies or food intolerance

Ages: 60 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-05-02 (Estimated); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-07-26 (Estimated)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass in kilograms (kg) | 3 months
  Appendicular skeletal muscle mass will be estimated using BIA in kilograms (kg). Prior to the assessment, participants will be screened to confirm they are not fitted with pacemakers. To ensure standardization, they will be instructed to remove footwear, socks, and any heavy accessories, as well as to empty their pockets and bladder. During the procedure, participants will be positioned at the center of the platform, standing upright with eyes forward while firmly holding the electrodes until the measurement is completed. BIA is selected for its simplicity, non-invasive nature, and suitability for field settings. Nevertheless, as hydration status can influence the readings, bladder emptying will be emphasized as a precaution to reduce measurement variability.
Appendicular skeletal muscle index (ASMI) in kilograms per square meter (kg/m²) | 3 months
  ASMI in kilograms per square meter (kg/m²) will be obtained by dividing an individual's appendicular skeletal muscle mass by the square of their height. Low skeletal muscle mass, a key diagnostic component of sarcopenia, was defined according to the AWGS 2025 criteria as an ASMI <7.6 kg/m² for men aged 50-64, <7.0 kg/m² for men aged 65 and above, and <5.7 kg/m² for women.
Muscle strength in kilograms (kg) | 3 months
  Muscle strength will be assessed using handgrip dynamometry and recorded in kilograms (kg). Three consecutive measurements will be obtained from the dominant hand, and the highest value will be used for analysis. Handgrip strength is a validated measure of overall muscle strength and is commonly used to assess muscular weakness.
  Muscle weakness will be defined according to the AWGS 2025 criteria. Low handgrip strength is defined as <34 kg for men aged 50-64 years, <28 kg for men aged ≥65 years, <20 kg for women aged 50-64 years, and <18 kg for women aged ≥65 years. Participants with handgrip strength below these sex- and age-specific thresholds will be classified as having muscle weakness.
  Muscle weakness identified by handgrip dynamometry will be used to operationalize the weakness component of the FFP and the muscle strength criterion within the AWGS sarcopenia framework.
Height in centimetres (cm) | 3 months
  Participants' height will not be obtained through direct standing height but will instead be estimated from arm span length, which is regarded as a more accurate indicator for older adults due to progressive reductions in height with ageing. Arm span refers to the distance measured between the tips of the middle fingers when both arms are fully stretched out to the sides. For the measurement procedure, each participant will be asked to stand upright against a wall with their back straight and arms extended horizontally at shoulder level. Measurements will be taken three times using a standardized metal measuring tape, and the average will be used for analysis. Predictive equations developed for Malaysian older adults will then be applied: for men, Height = [0.681 × arm span (cm)] + 47.56; and for women, Height = [0.851 × arm span (cm)] + 18.78.
Body weight in kilograms (kg) | 3 months
  Body weight will be assessed using BIA with the InBody 270 device. Prior to the assessment, participants will be screened to confirm they are not fitted with pacemakers. To ensure standardization, they will be instructed to remove footwear, socks, and any heavy accessories, as well as to empty their pockets and bladder. During the procedure, participants will be positioned at the center of the platform, standing upright with eyes forward.
Body mass index (BMI) in kilograms per square meter (kg/m²) | 3 months
  BMI, which will be obtained by dividing body weight in kilograms by the square of height in meters (kg/m²). Among older adults, an optimal BMI is expected to fall between 24 and 27 kg/m². Readings below 24 kg/m² will indicate underweight status, while values exceeding 27 kg/m² will reflect overweight conditions.
Body fat percentage in percentage (%) | 3 months
  Body fat percentage will be measured using BIA. Male participants presenting with 25% or more body fat will be identified as obese, while those below this level will be considered non-obese. For females, obesity will be defined at 35% or higher body fat, with measurements under this threshold reflecting a non-obese status.
Waist circumference in centimetres (cm) | 3 months
  Waist circumference of the participants will be measured using a metal measuring tape. Male participants with a waist circumference of 90 cm or above will be categorized as having abdominal obesity, while those with measurements below 90 cm will be considered non-abdominally obese. For female participants, abdominal obesity will be defined as a waist circumference of 80 cm or greater, with values under 80 cm classified as non-abdominally obese.
Calf circumference in centimetres (cm) | 3 months
  Calf circumference will be assessed using a metal measuring tape. The measurement will be taken at the widest part of the calf, ensuring the tape is positioned horizontally and parallel to the floor. During the assessment, participants will be seated with knees and ankles flexed at 90°, feet resting flat on the ground. To ensure precision, the tape will be placed directly on the skin without clothing interference.
Cognitive performance | 3 months
  Cognitive frailty will be evaluated based on the presence of both cognitive impairment and physical frailty. Cognitive performance will be assessed using the MoCA, which is scored from 0 to 30, with higher scores indicating better cognitive function. For classification purposes, MoCA scores will be interpreted as follows: Normal cognition: 26-30; MCI: 18-25; Moderate to severe impairment: ≤17
  Participants who demonstrate mild cognitive impairment (MoCA score 18-25) in combination with pre-frailty or frailty (FFP score ≥2) will be classified as having cognitive frailty.
Malaysian-MIND diet (MY-MINDD) score | 3 months
  Baseline and follow-up 7-day diet histories will be collected, and adherence to the MY-MINDD will be evaluated using the MY-MINDD score, a tool specifically developed for Malaysian older adults. Dietary intake will be assessed based on 11 food groups: whole grains, green leafy vegetables, other vegetables, flavonoid-rich fruits, deep-sea fish (non-fried), poultry (non-fried), legumes and soy products, desserts, sweetened kuih and beverages, red meat, fried/fast foods, and butter/margarine. Each group will be scored according to intake frequency and serving sizes (0, 0.5, or 1). The total score will be obtained by summing all components, with a maximum of 11 points, which is a modified version of the original MIND diet score (15 points). An increased score will denote stronger compliance with the MY-MINDD dietary guidelines.
Unintentional Weight Loss in kilogram (kg) | 3 months
  Unintentional weight loss will be assessed by self-report. Participants will be asked whether they have experienced an unintentional weight loss of >10 kg of their body weight within the past 12 months. Participants meeting this criterion will be classified as fulfilling the weight loss component of the FFP.
Exhaustion | 3 months
  Exhaustion will be assessed using two items from the Center for Epidemiologic Studies Depression Scale (CES-D):
  "I felt that everything I did was an effort," and "I could not get going."
  Participants reporting either symptom for ≥3 days per week during the past week will be classified as having exhaustion, thereby fulfilling the exhaustion component of the FFP.
Physical Performance in seconds (s) | 3 months
  Physical performance will be assessed using the 5t-CST. Participants will be instructed to stand up and sit down five times as quickly as possible from a standard chair without using their arms. The total time to complete five repetitions will be recorded in seconds.
  Slowness will be defined based on established cut-off values for the 5t-CST. Participants with performance times exceeding the specified threshold will be classified as fulfilling the slowness component of the FFP.
Physical Activity Score | 3 months
  Physical activity level will be assessed using a validated PASE questionnaire. The PASE assesses the frequency and duration of leisure-time, household, and occupational physical activities performed over the previous 7 days. Weekly energy expenditure will be calculated and expressed in kilocalories per week (kcal/week).
  Low physical activity will be defined according to sex-specific cut-off values consistent with the FFP. Participants with weekly energy expenditure below the specified thresholds will be classified as fulfilling the low physical activity component of the Fried Frailty Phenotype.
Frailty | 3 months
  Frailty will be assessed using the FFP, a validated multidimensional construct comprising five components: unintentional weight loss, exhaustion, weakness, slowness, and low physical activity. Each component will be assessed according to standardized criteria.
  Participants will be classified based on the total number of criteria met: robust (0 criteria), pre-frail (1-2 criteria), and frail (≥3 criteria). Frailty status will be used as a categorical outcome measure in the present study.

SECONDARY OUTCOMES:
Incremental Cost-Effectiveness Ratio (ICER) | 3 months
  Direct costs for the intervention group, including food ingredients, packaging, transportation, and staff wages, will be calculated. Effectiveness will be measured using quality of life (QoL) and medical costs.
  Quality of life will be evaluated using CASP-19 questionnaire which consists of 19 items. Scores range from 0 to 57, with higher scores indicating better quality of life.
  Medical costs, including outpatient visits, hospitalization, complementary and alternative medicine (CAM) use, and post-hospitalization rehabilitation, will be self-reported by participants throughout the three-month intervention.
  The incremental cost-effectiveness ratio (ICER), representing the additional cost required to achieve one additional unit of health benefit, will be calculated as the difference in costs between the intervention and control groups divided by the difference in outcomes (QoL or medical costs) between the two groups.
Brain-Derived Neurotrophic Factor (BDNF) in picograms per milliliter (pg/mL) | 3 months
  Venous blood samples will be collected from participants by trained personnel using standard aseptic procedures. The samples will be processed to obtain serum and stored appropriately before being transported to an accredited laboratory for analysis. Quantification of brain-derived neurotrophic factor (BDNF) will be conducted by laboratory experts using a commercially available enzyme-linked immunosorbent assay (ELISA) kit to ensure accuracy and reliability of the results.
6-item USDA Household Food Security Survey Module (HFSSM) score | 3 months
  Food security will be evaluated using the validated 6-item USDA Household Food Security Survey Module (HFSSM), which includes six questions. Responses of "often" or "sometimes" to HH3 and HH4, as well as "yes" to AD1, AD2, and AD3, will be coded as affirmative. For AD1a, responses of "almost every month" or "some months but not every month" will also be considered affirmative. Each affirmative response will be awarded one point, and the total will represent the raw score. A raw score of 0-1 will indicate high or marginal food security, 2-4 will indicate low food security, and 5-6 will indicate very low food security. In this study, both English and Malay versions of the 6-item HFSSM will be administered.
Depressive Symptoms | 3 months
  Depressive symptoms will be assessed using the 15-item Geriatric Depression Scale (GDS-15), a validated self-report screening tool for depressive symptoms in older adults. The GDS-15 evaluates mood and affect based on yes/no responses reflecting symptoms experienced over the past week.
  Total scores range from 0 to 15, with higher scores indicating greater depressive symptom severity. A score of ≥5 will be used to indicate the presence of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yoke Mun Prof. Dr. Chan, Ph.D(Community Nutrition)(UPM), Principal Investigator — Universiti Putra Malaysia
Locations (2):
- Malaysia (2):
  - Perumahan Awam (PA) Loke Yew, Kuala Lumpur
  - Project Perumahan Rakyat (PPR) Seri Alam Fasa 2, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No